CLINICAL TRIAL: NCT03019653
Title: A Phase Ib, Double-Blind, Placebo-Controlled, Single-site Trial to Determine the Safety and Efficacy of a Novel Renal-Specific Peptide, ANX-042, in Enhancing GFR Without Significant Hypotension in Human Cardiorenal Syndrome (CRS): ANX-042 Aim #1
Brief Title: Safety and Efficacy of ANX-042 in Human Cardiorenal Syndrome
Acronym: ANX-042 Aim 1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Paul M. McKie, M.D., PI, Mayo Clinic
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 16-001847; R01HL084155-06A1 (NIH)
Record Dates: First submitted 2017-01-11; First posted 2017-01-12 (Estimated); Last update posted 2024-11-15 (Actual); Status verified 2024-11

CONDITIONS: Heart Failure; Cardiorenal Disease; Renal Disfunction
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | US Export: No

ARMS (2):
- ANX-042 first, then Placebo (Active Comparator): In the first intervention period the subjects will receive an infusion of ANX-042. There will be a 3 week washout period. In the second intervention period, the subjects will receive an infusion of placebo
  Interventions: Drug: ANX-042; Drug: Placebo
- Placebo first, then ANX-042 (Active Comparator): In the first intervention period the subjects will receive placebo. There will be a 3 week washout period. In the second intervention period, the subjects will receive an infusion of ANX-042.
  Interventions: Drug: ANX-042; Drug: Placebo

INTERVENTIONS:
Drug: ANX-042 — The first 20 subjects will receive a dose 0.003 µg/kg/min by infusion, the next 20 subjects will receive a dose of 0.006 µg/kg/min, then the next 20 subjects will receive 0.01 µg/kg/min.
Drug: Placebo — The pharmacy created a placebo for this study is sterile Dextrose (5%) solution (D5W) 0.9% Sodium Chloride for intravenous administration to match study drug.

SUMMARY:
The purpose of this study is to look at kidney function and hormonal function in patients with a history of heart failure and kidney dysfunction, and to see how the use of a new drug, ANX-042, affects those functions.

DETAILED DESCRIPTION:
Subjects will have a choice of admitting the night prior to renal clearance study day or the day of. Subjects will admit (fasting) to the Clinical Research and Trials Unit, after 3 weeks of diet compliance, the morning of the first renal clearance study day. They will avoid taking any sulfa containing medications and Probenecid for 72 hours prior to Visit Two and Visit Three. They will complete a 24-hour urine collection which will be assessed for creatinine clearance, microalbumin and sodium concentration and excretion. A pregnancy test will be performed, if necessary. Their first urine void after admitting will be collected for protein analysis. Brief physical exam (same as at Visit 1) will be performed by a qualified Study Team Member. Their usual morning dose of medications will be held until given initial water load prior to start of renal clearance infusion. Echocardiogram to determine systolic, diastolic function and cardiac output will be performed prior to the start of study drug infusion. A bladder ultrasound will be performed after their first void. If subject is unable to sufficiently empty their bladder, a urinary catheter will be placed with their permission. The subjects will be placed in the supine position for 1 hour. During the first 15 minutes, two standard intravenous (IV) catheters will be placed (one in each arm). One catheter will be used for infusion and the other (in the contralateral arm) for blood sampling. Subjects will be asked to drink 5 mL/Kg of water initially and then drink an amount equal to the urine output, and blood drawn, after each clearance period to ensure sufficient urinary flow. A priming dose (calculated according to body size) of iothalamate (0.06 mg/Kg) to measure glomerular filtration rate (GFR) will be infused, followed by a constant rate IV sustaining dose (calculated according to estimated kidney function) of iothalamate to achieve steady-state plasma concentrations of 15 to 20 mg/L. The subjects will be asked to empty their bladder spontaneously at the end of each clearance period.

After an equilibration period of 45 minutes, urine and blood samples will be collected at 30-minutes to determine the baseline GFR and urinary sodium excretion (UNaV). Blood pressure will be measured at 20-minute intervals for the first 2 hours, then every 30 minutes, by using automatic blood pressure cuff. Heart rate will be continuously monitored by electrocardiography. Urinary samples for determination of volume, sodium, potassium, and iothalamate will be obtained at the end of each clearance period. Venous blood samples for iothalamate and sodium will be obtained at the middle of each clearance period. During the first clearance, venous blood samples for renin, aldosterone, angiotensin II, AnxA1, Atrial Natriuretic Peptide (ANP), Brain natriuretic peptide (BNP) and cGMP will be obtained and urine samples for Annexin A1(AnxA1) and cyclic guanosine monophosphate (cGMP) will also be obtained. Buffy coat from Ethylenediaminetetraacetic acid (EDTA) vacutainer tubes will be saved for possible future DNA analysis.

After the baseline renal clearance, subjects will be randomized to receive infusion of active study drug or placebo for 8 hours. The research pharmacist will prepare the study drug or placebo infusion, thus both the patients and investigators will be blinded. Renal clearance and blood draws will be carried out every 2 hours during the infusion as described above (4 times), and blood draw for assays at the end of 4 and 8 hours infusion as listed above. Another echocardiogram will be repeated after 4 hour of drug infusion. Subjects will be given 3 meals throughout the day. Dismissal will occur after one hour of post-infusion monitoring.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular ejection fraction of equal or less than 40% assessed by echocardiography, nuclear scan, MRI or left ventriculogram within the past 48 months. If assessment is greater than 12 months old, hand-held echocardiogram (ECHO) determination will be performed at consent visit once enrolled.
* Stable New York Heart Association (NYHA) class II and III symptoms as defined by: no change in NYHA symptoms over the past 3 months, on stable doses of furosemide, angiotensin-converting enzyme (ACE) inhibitor or angiotensin II type 1 (AT1) blocker, beta blocker, or aldosterone antagonist over the last 4 weeks and no episode of decompensated Congestive Heart Failure (CHF) over the past 6 months.
* Calculated creatinine clearance of equal or less than 89 ml/min and greater than 20 ml/min, using the Modification of Diet in Renal Disease (MDRD) formula assessed within the past 48 months and a confirmatory calculated creatinine clearance equal or less than 89 ml/min and greater than 20 ml/min at the time of enrollment.
* Digoxin, antiarrhythmic medications and other vasodilators will be allowed; however, all medications must be at stable doses 4 weeks prior to enrollment. Subjects taking non-steroidal anti-inflammatory drugs (NSAIDs), except aspirin, will not be able to increase their medication dose for the duration of the study.

Exclusion Criteria:

* Prior diagnosis of intrinsic renal diseases, such as glomerular nephritis or polycystic kidney disease, including renal artery stenosis of > 50% (unless revascularized)
* Peritoneal or hemodialysis within 90 days or anticipation that dialysis or ultrafiltration of any form will be required during the study period
* Hospitalization for decompensated CHF during the past 6 months
* Myocardial infarction within 6 months of screening
* Unstable angina within 6 months of screening, or any evidence of acute myocardial ischemia
* Significant valvular stenosis (greater than moderate in severity) , hypertrophic, restrictive or obstructive cardiomyopathy, constrictive pericarditis, primary pulmonary hypertension, or biopsy proven active myocarditis
* Severe congenital heart diseases
* Sustained ventricular tachycardia or ventricular fibrillation within 14 days of screening
* Second or third degree heart block without a permanent cardiac pacemaker
* Stroke within 3 months of screening, or other evidence of significantly compromised central nervous system (CNS) perfusion
* Alanine transaminase (ALT) >2 times the upper limit of normal
* Serum sodium of < 125 milliequivalent/dL (mEq/dL) or > 160 mEq/dL
* Serum potassium of < 3.0 mEq/dL or > 5.7 mEq/dL
* Hemoglobin < 8.5 gm/dl
* Other acute or chronic medical conditions or laboratory abnormality which may increase the risks associated with study participation or may interfere with interpretation of the data
* Have received an investigational drug within 1 month prior to dosing
* Patients with an allergy to iodine
* Female subject who is pregnant or breastfeeding
* In the opinion of the investigator, is unlikely to comply with the study protocol or is unsuitable for any reasons
* Documented systolic blood pressure less than 90 mmHg at consent visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2024-09-13 (Actual); Study Completion 2024-09-13 (Actual)

PRIMARY OUTCOMES:
Change in Glomerular Filtration Rate | baseline to 3 weeks

SECONDARY OUTCOMES:
Change in Sodium Excretion | baseline to 3 weeks
Change in Urine Flow | baseline to 3 weeks
Change in Blood Pressure | baseline to 3 weeks
Change in Renin-angiotensin-aldosterone system (RAAS) | baseline to 3 weeks
Change in Urine Annexin A1 (AnxA1) Protein Levels | baseline to 3 weeks
Number of Subjects with Hypotension | 3 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Paul M McKie, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No